CLINICAL TRIAL: NCT03144154
Title: Impact of an Intervention Combining Self-care and Hypnosis on the Well-being of Cancer Patients and Their Partners
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Liege (Other)
Collaborators: King Baudouin Foundation (Other); Jules Bordet Institute (Other); Fonds National de la Recherche Scientifique (Other)
Responsible Party: Principal Investigator, Isabelle Bragard, PhD, University of Liege
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Onco-Hypn-Fatigue
Record Dates: First submitted 2017-05-01; First posted 2017-05-08 (Actual); Last update posted 2020-09-28 (Actual); Status verified 2020-09

CONDITIONS: Non-Metastatic Neoplasm
Keywords: Cancer; Fatigue; Hypnosis; Self-hypnosis; Self-care; Emotional distress; Cancer survivors
MeSH Terms: conditions — Neoplasms; Fatigue | interventions — Hypnosis; Self Care

STUDY DESIGN:
Intervention Model Description: Participants are randomized into 2 groups: the experimental group receives the intervention immediately while the control group only receives usual care. When the control group has received the intervention and that evaluations have been done for all participants, the control group will receive the intervention (randomized controlled trial).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group : Hypnosis-based intervention (Experimental): Groupal intervention combining self-care techniques and self-hypnosis exercises
  Interventions: Behavioral: Self-hypnosis + Self-care
- Control group : Usual care (No Intervention): Control group receiving usual care but not the intervention

INTERVENTIONS:
Behavioral: Self-hypnosis + Self-care — Our groupal intervention is divided into 8 weekly 2-hour sessions in which one self-hypnosis exercise is proposed to participants. Self-care techniques are also discussed (knowing our own needs, self-respect, assertiveness, coping with ruminations...) and homework assignments are proposed to participants, in order to foster positive change.
  Arms: Experimental group : Hypnosis-based intervention

SUMMARY:
Hypnosis-based interventions are starting to be tested in order to improve emotional distress and fatigue of cancer patients. However, most of these studies only include breast cancer patients and do no measure long-term effects of such interventions.

Our randomized controlled trial aims to propose to 116 post-treatment cancer patients (all tumour localisations accepted) an 8-week groupal intervention combining hypnosis and self-care techniques.

Primary outcomes (emotion regulation, emotional distress, fatigue) and secondary outcomes (sleep difficulties, fear of recurrence, attentional bias, conjugal communication) will be investigated at 3 measurement times: before the intervention (T1), 3 months later (T2 - right after the intervention of the experimental group, and right before the intervention of the control group) and again 3 months later (T3 - after the intervention of the control group). Some questionnaires, two relaxation tasks, an attentional task, an actigraph and a smartphone application will be used to collect data. The indirect impact of the intervention on participants' partners will also be measured by questionnaires (emotional distress, conjugal communication).

Data collection has started on March 2017. Our results should bring new knowledge about the efficacy of an hypnosis-based intervention to improve fatigue and well-being in cancer patients, which are often under-diagnosed and under-treated, but also about the indirect efficacy to improve partners' well-being. Those results might contribute to spread this kind of inexpensive intervention in oncology settings.

ELIGIBILITY:
Inclusion criteria are:

1. age 18 years or older;
2. Fluency in French;
3. Having received a diagnosis of non-metastatic cancer (all tumour localisations accepted).
4. Having completed all active treatments for no more than a year (surgery, chemotherapy and radiotherapy).
5. Not being in relapse at the time of inclusion
6. Exhibiting some difficulties as established by responses of at least 4 out of 10 on 1 of the 6 chosen items of the Edmonton Symptom Evaluation Scale (Chang, Hwang, & Feuerman, 2000): physical fatigue, moral fatigue, depression, anxiety, fear of recurrence or ruminations).
7. Wishing to receive help in order to improve the difficulties identified.

Exclusion Criteria:

Psychiatric disorders, such as dementia, psychosis or delirium, that do not allow to participate in a group intervention or to complete the evaluations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2017-02-13 (Actual); Primary Completion 2019-10-20 (Actual); Study Completion 2020-09-18 (Actual)

PRIMARY OUTCOMES:
Change in Cancer-Related Fatigue | T1 (before the intervention), T2 (right after the intervention), T3 (3.5 months follow-up)
  A sense of tiredness or exhaustion linked with cancer and its treatments, that is not alleviated by sleep. It will be measured with the Multidimensional Fatigue Inventory (MFI-20) and the Insomnia Severity Index (ISI).
Change in emotional distress | T1 (before the intervention), T2 (right after the intervention), T3 (3.5 months follow-up)
  Anxiety + Depression, measured with the Hospital Anxiety and Depression Scale (HADS)

SECONDARY OUTCOMES:
Change in fear of recurrence | T1 (before the intervention), T2 (right after the intervention), T3 (3.5 months follow-up)
  Fear that cancer could return. Measured with the Fear of Cancer Recurence Inventory
Change in emotion regulation | T1 (before the intervention), T2 (right after the intervention), T3 (3.5 months follow-up)
  The way people deal with their emotions. Measured with one questionnaire (Cognitive Emotion Regulation Questionnaire) and a smartphone application asking participants about their daily emotion and how they deal with it. The application is used during 9 days at each measurement time.
Change in attentional bias towards threat | T1 (before the intervention), T2 (right after the intervention), T3 (3.5 months follow-up)
  Attentional bias toward emotional information especially negative ones. It is linked with anxiety and will be measured by an computerized task.
Change in the quality of the conjugal relationship | T1 (before the intervention), T2 (right after the intervention), T3 (3.5 months follow-up)
  Communication about cancer and dyadic coping, measured with questionnaires (Couples' Illness Communication Scale ; Dyadic Coping Inventory). The two partners will complete these questionnaires.
Change in partners' well-being | - Couples' Illness Communication Scale (CICS) (Arden-Close et al., 2010) Dyadic Coping Inventory (DCI)
  Anxiety and depression of the partners, measured with the HADS.

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Elisabeth Faymonville, Study Director — CHU de Liège - Université de Liège
Locations (1):
- University Hospital of Liege, Liège, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Baussard L, Ernst M, Diep A, Jerusalem G, Vanhaudenhuyse A, Marie N, Bragard I, Faymonville ME, Gosseries O, Gregoire C. Network Analyses Applied to the Dimensions of Cancer-Related Fatigue in Women With Breast Cancer. Cancer Med. 2024 Oct;13(19):e70268. doi: 10.1002/cam4.70268. PMID 39387227
- [Derived] Gregoire C, Faymonville ME, Vanhaudenhuyse A, Jerusalem G, Monseur J, Bragard I. A Group Intervention Combining Self-Hypnosis and Self-Care in Oncology: Implementation in Daily Life and Perceived Usefulness. Int J Clin Exp Hypn. 2023 Oct-Dec;71(4):313-337. doi: 10.1080/00207144.2023.2249044. Epub 2023 Sep 8. PMID 37682079
- [Derived] Gregoire C, Faymonville ME, Vanhaudenhuyse A, Jerusalem G, Willems S, Bragard I. Randomized, Controlled Trial of an Intervention Combining Self-Care and Self-Hypnosis on Fatigue, Sleep, and Emotional Distress in Posttreatment Cancer Patients: 1-Year Follow-Up. Int J Clin Exp Hypn. 2022 Apr-Jun;70(2):136-155. doi: 10.1080/00207144.2022.2049973. Epub 2022 Mar 28. PMID 35344461
- [Derived] Gregoire C, Faymonville ME, Vanhaudenhuyse A, Jerusalem G, Willems S, Bragard I. Randomized controlled trial of a group intervention combining self-hypnosis and self-care: secondary results on self-esteem, emotional distress and regulation, and mindfulness in post-treatment cancer patients. Qual Life Res. 2021 Feb;30(2):425-436. doi: 10.1007/s11136-020-02655-7. Epub 2020 Oct 6. PMID 33025372
- [Derived] Gregoire C, Faymonville ME, Vanhaudenhuyse A, Charland-Verville V, Jerusalem G, Willems S, Bragard I. Effects of an intervention combining self-care and self-hypnosis on fatigue and associated symptoms in post-treatment cancer patients: A randomized-controlled trial. Psychooncology. 2020 Jul;29(7):1165-1173. doi: 10.1002/pon.5395. Epub 2020 Apr 24. PMID 32297396
- [Derived] Gregoire C, Faymonville ME, Vanhaudenhuyse A, Charland-Verville V, Jerusalem G, Bragard I. Randomized controlled trial of an 8-week intervention combining self-care and hypnosis for post-treatment cancer patients: study protocol. BMC Cancer. 2018 Nov 15;18(1):1113. doi: 10.1186/s12885-018-5046-6. PMID 30442120